CLINICAL TRIAL: NCT05644834
Title: IGHID 12227 - Pilot Mobile Medical Unit Study for I'm Fully Empowered4Her (IFE4Her) Intervention on HIV Pre-Exposure Prophylaxis (PrEP) Uptake by Women Living in Durham Housing Authority - Affiliated Communities (IFE4Her Pilot Study)
Brief Title: Pilot Mobile Medical Unit Study for I'm Fully Empowered4Her
Acronym: IFE4Her
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Gilead Sciences (Industry); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-1570
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: HIV Prevention; Pre-exposure Prophylaxis; PrEP; Prevention; Women's Health; Mobile Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Medical Unit (Experimental): Participants utilizing the mobile medical unit will be offered an appointment with a university system healthcare provider to receive blood pressure check, blood glucose check, HIV testing and/or Pre-exposure Prophylaxis (PrEP) consultation.
  Interventions: Other: I'm Fully Empowered for Her (IFE4Her)

INTERVENTIONS:
Other: I'm Fully Empowered for Her (IFE4Her) — IFE4Her consists of 2 key components: 1) An awareness-raising messaging campaign with messages about PrEP that includes posters and Peer Networkers; and 2) access via a mobile medical unit outreach delivery model linking women in public housing to care from the PrEP providers of a university healthcare system and other complementary screening services (i.e., blood pressure, blood glucose monitoring, and HIV testing).

SUMMARY:
The overarching objective for the pilot study is to test the feasibility of using a mobile medical unit as a delivery mode combined with enhanced Pre-exposure Prophylaxis (PrEP) messaging to increase awareness of PrEP and access to PrEP medical services among women living in public housing.

DETAILED DESCRIPTION:
This is a single arm feasibility study with 3-month follow-up.

African American cisgender women in the South are disproportionately affected by HIV infection yet have inequitable access to Pre-exposure Prophylaxis (PrEP). To promote equitable use of PrEP by women living in low-income housing in Durham, North Carolina (NC) (the vast majority of whom are African American), the investigators aim to conduct a formative study to develop and refine a scalable PrEP delivery approach which addresses the two key barriers of access and awareness. In this pilot study the investigators will test the feasibility of the delivery mode and features of a community outreach PrEP mobile unit and provide Peer Networkers and PrEP messaging tailored to women living in public housing.

The objectives of the study are to evaluate the feasibility of delivering the IFE4Her intervention in public housing communities. The IFE4Her intervention consists of: 1) a communication campaign including enhanced PrEP messaging and peer networker communication; 2) A mobile PrEP clinic. Assessments will include a satisfaction survey for participants receiving services in the mobile clinic, service records, follow-up in-depth interviews at 3 months, and chart review at 6 months to assess 3-month outcomes.

Study Duration Each participant's study duration will depend upon the study activities they elect to engage in. Each subject's participation in the anonymous survey will last approximately 10 minutes immediately after their medical visit. Each subject's participation in the follow-up interview which will take place approximately 3 months after the mobile medical visit and will last approximately one hour. Medical record data (specifically follow up visit participation and prescription completion as described in detail below) will be collected after the 3 month visit but up to 6 months after participation in the initial medical visit.

The entire pilot study is expected to last up to 2 years.

Intervention Description

1. Communication campaign

   1. Communication Materials - PrEP Posters and Infographics that provide information about PrEP for women, and materials on complementary health services including hypertension screening, blood glucose screening, and HIV-testing.
   2. Peer Networker Information Dissemination - Trained Peer Networkers will disseminate information about PrEP, complementary women's health issues, and the mobile medical unit through distribution of communication materials and in-person communication.
2. Mobile Medical Unit All study-related clinical services will occur in a safe, confidential, and private space in a mobile medical unit. The mobile medical unit will offer the following services: blood pressure checks, blood glucose monitoring, rapid HIV antibody testing, and for those interested, PrEP consultation and clinical assessment and care as indicated. These services will be provided by university health care system clinicians. Participants receiving PrEP will be receive follow-up care in the university health care system.

Of note, no study drug is being tested. The PrEP medication emtricitabine/tenofovir disoproxil fumarate (trade name Truvada®) that providers will write prescriptions for is the only medication currently approved for women. It is very well tolerated and taken once daily. Truvada prescriptions will be provided in accordance with standard clinical care. These decisions are not protocol/study-driven and not an intervention being studied by the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Identify as female
* Currently reside in Durham Housing Authority (DHA) housing

Exclusion Criteria:

* Currently on PrEP or Post-Exposure Prophylaxis (PEP)
* HIV-positive
* Being Male Gender
* Altered mental status precluding participant to provide informed consent
* Currently Pregnant or Trying to get Pregnant or Lactating.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female
Enrollment: 35 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability - Mean Score of Satisfaction Questionnaire (range 1-5 with higher scores meaning greater satisfaction) | Immediately post-mobile medical unit visit (assessed an average of 10 minutes post mobile medical unit visit)
  Perceived satisfaction with the intervention as assessed through survey items
Intervention Acceptability - Number of Completed PrEP Consultations | Immediately post-mobile medical unit visit (assessed an average of 10 minutes post mobile medical unit visit)
  Number of mobile clinic clients completing a PrEP consultation with a study provider as recorded by study staff in service records
Intervention Acceptability Assessed Qualitatively | 3 months
  Perceived acceptability of the intervention as assessed in qualitative in-depth interviews with mobile clinic clients
  To gain deeper insights about the perceived acceptability of the intervention the investigators will ask participants in in-depth interviews about how they about different aspects of the intervention, including services provided and their delivery. Acceptability will be defined as a positive rating (and reason for that rating) of participant satisfaction with each aspect of the intervention.

SECONDARY OUTCOMES:
PrEP uptake - Number of PrEP Prescriptions Written in the Mobile Clinic | Immediately post-mobile medical unit visit (assessed an average of 10 minutes post mobile medical unit visit)
  PrEP uptake, assessed as PrEP prescriptions written for women in the target population from the mobile PrEP unit evaluated through service records
PrEP persistence -Proportion of Participants Receiving a PrEP Prescription Who Completed a Follow-Up visit and Received a Follow-Up PrEP Prescription | 3 months
  Persistence in PrEP care, assessed via chart review of follow-up appointments and prescriptions documented in Duke clinic records as the proportion of participants who received a PrEP prescription and completed a follow-up visit and received a follow-up PrEP prescription at 3 months (assessed retrospectively at 6 months).
PrEP Consultation Requests - Number of PrEP Appointments Requested | Baseline
  Number of mobile unit PrEP consultations (either scheduled or walk-in) requested as recorded in study tracking records and service logs.
PrEP Consultation Uptake - Number of PrEP Consultations Completed | Immediately post-mobile medical unit visit (assessed an average of 10 minutes post mobile medical unit visit)
  Number of mobile unit PrEP consultations (either scheduled or walk-in) completed as recorded in mobile unit service logs

CONTACTS AND LOCATIONS:
Overall Officials: Carol Golin, MD, Principal Investigator — UNC-Chapel Hill; Lauren Hill, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.